CLINICAL TRIAL: NCT03948061
Title: Cardiometabolic Effects of Sweet Cherry Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Washington State Fruit Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FL108
Record Dates: First submitted 2019-04-25; First posted 2019-05-13 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: cherries; inflammatory disease; chronic stress
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cherry juice followed by placebo (Experimental): Sweet cherry juice concentrate will be consumed twice daily for 6 weeks, followed by consumption of placebo beverage twice daily for 6 weeks.
  Interventions: Other: Cherry juice; Other: Placebo beverage
- Placebo beverage followed by cherry juice (Experimental): Placebo beverage will be consumed twice daily for 6 weeks, followed by consumption of sweet cherry juice concentrate twice daily for 6 weeks.
  Interventions: Other: Cherry juice; Other: Placebo beverage

INTERVENTIONS:
Other: Cherry juice — FruitSmart® Cherry Concentrate: Dark Sweet Cherry Juice Concentrate produced from dark sweet cherries to retain the characteristic color and flavor of the whole fruit.
Other: Placebo beverage — Cherry flavored placebo beverage prepared from commercially available cherry syrup with food coloring and thickener to match the color and viscosity of the cherry concentrate.

SUMMARY:
This study aims to determine the effects of consuming sweet cherry juice on cardiovascular function, glucose regulation, and lipid status in overweight human subjects. The investigators hypothesize that sweet cherry juice consumption will improve metabolic and physiological status in overweight persons compared to a placebo.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, cross-over study lasting 14 weeks and including 1 week for screening/enrollment, 1 week baseline assessment, and two intervention periods of 6 weeks each for the cherry juice and placebo interventions. Two test visits, 3 to 7 days apart, will occur before the start of intervention (baseline, or week 0) and then at weeks 6 and 12. Participants will be randomized to consume either the cherry juice or placebo beverage first, and will cross over to the alternate intervention immediately following the end of the first 6 weeks. Test Visit 1 will include measures of blood pressure, vascular tone, liver fat and stiffness, post-prandial metabolic response to the study beverage, cardiovascular activity and function, and nervous system control of cardiovascular activity and tone. Acute effects of study beverages will be measured, as will the chronic effects of study beverage consumption after 6 weeks. At Test Visit 2, participants will take a standard 75 gram oral glucose tolerance test (OGTT). Participants will be equipped with physiological monitoring devices, which will monitor cardiovascular activity and function and nervous system control of cardiovascular activity and tone, and continuously measure blood pressure. A series of cognitive function tasks will be administered, and a mental stress test will be conducted. The Test Visit 1 and 2 will be repeated at week 6 and week 12 following each intervention with cherry juice or the placebo beverage.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 - 65 years
* Post-menopausal women aged 45 - 65 years
* Body Mass Index ≥25 and <40 kg/m2
* Systolic blood pressure >120 and <140 mmHg or diastolic blood pressure >80 and <90 mmHg

Exclusion Criteria:

* Diagnosed metabolic disorder
* Diabetes mellitus
* Thyroid disease
* Cardiovascular disease
* Poly-cystic ovary syndrome
* Vasoconstrictive diseases (e.g. Raynaud's phenomenon or Raynaud's disease)
* Digestive disorder (e.g. Crohn's, irritable bowel syndrome, colitis)
* History of gastrointestinal surgery affecting digestion and/or absorption
* Use of medications for hypertension, hyperlipidemia, glycemic control, or weight loss
* Use of medications such as steroids, statins, or non-steroidal anti-inflammatory agents
* Routine use of over-the-counter medications
* Weight change >5% in the past 6 months
* Performing exercise greater than 60 minutes/day
* Presence of a pacemaker or other internal electronic device controlling rhythm or pacing of heart excludes participant from MindWare procedure
* Presence of atrial fibrillation or other arrhythmia excludes participant from MindWare procedure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Week 0, 6 and 12
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg
Change in diastolic blood pressure | Week 0, 6 and 12
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg
Change in mean arterial blood pressure | Week 0, 6 and 12
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg
Change in heart rate variability | Week 0, 6 and 12
  Heart rate variability (HRV) assessed using a mobile device via ECG in millivolts
Change in cardiac parasympathetic control | Week 0, 6 and 12
  Assessed using impedance cardiography (ICG) and ECG
Change in electrical activity of heartbeat | Week 0, 6 and 12
  Assessed using electrocardiogram (ECG)

SECONDARY OUTCOMES:
Change in vascular function | Week 0, 6 and 12
  Peripheral arterial tone (PAT) determined using the EndoPAT expressed as the reactive hyperemia index (RHI)
Change in liver stiffness | Week 0, 6 and 12
  Liver stiffness assessed from the shear wave speed with pulse echo ultrasound using the Fibroscan®
Change in liver fat | Week 0, 6 and 12
  Liver fat assessed from the Controlled Attenuation Parameter (CAP) computed from the liver stiffness measurement using the Fibroscan®
Change in executive function | Week 0, 6 and 12
  Assessed using Cambridge Gambling Task (CGT), from Cambridge Neuropsychological Test Automated Battery (CANTAB)
Change in attentive function | Week 0, 6 and 12
  Assessed using Stop Signal Task (STT) from CANTAB
Change in multitasking | Week 0, 6 and 12
  Assessed using Multitasking Test (MTT) from CANTAB
Change in psycho-motor speed | Week 0, 6 and 12
  Assessed using Reaction Time (RTI) task from CANTAB
Change in spatial memory | Week 0, 6 and 12
  Assessed using Spatial Working Memory (SWM) task from CANTAB
Change in verbal memory | Week 0, 6 and 12
  Assessed using Verbal Recognition Memory (VRM) task from CANTAB
Change in social cognition | Week 0, 6 and 12
  Assessed using Emotional Recognition task (ERT) from CANTAB
Change in peripheral insulin resistance (IR) | Week 0, 6 and 12
  Measured by Matsuda's sensitivity index
Change in hepatic insulin resistance (IR) | Week 0, 6 and 12
  Measured by homeostasis model assessment (HOMA)
Change in salivary cortisol in response to glucose tolerance test | prior to and 120 minutes after glucose tolerance test
  Salivary cortisol measured by enzyme-linked immunoassay in nmol/liter
Change in salivary cortisol in response to stress | prior to and 30, 60, 90 and 120 minutes after challenging task
  Salivary cortisol measured by enzyme-linked immunoassay in nmol/liter
Change in body weight | Week 0, 6 and 12
  Measured in kg
Change in waist circumference | Week 0, 6 and 12
  Measured in cm
Change in activity level | Week 0, 6 and 12
  Measured by Stanford Brief Physical Activity questionnaire. Scale is categorical for two subscales: work physical activity and leisure time activity.
Change in mitochondrial respiration | Week 0, 6 and 12
  Cellular bioenergetics measured as oxygen consumption rate (OCR)
Change in cardiovascular related biomarkers | Week 0, 6 and 12
  Quantitative immunoassay of human cardiovascular biomarkers on a multi-analyte profile
Change in inflammation related biomarkers | Week 0, 6 and 12
  Quantitative immunoassay of human inflammation biomarkers on a multi-analyte profile
Change in neurological related biomarkers | Week 0, 6 and 12
  Quantitative immunoassay of human neurological biomarkers on a multi-analyte profile
Change in perceived stress | Week 0, 6 and 12
  Perceived stress measured using the Perceived stress scale (PSS). Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Responses for individual questions are summed to a total score.
Change in chronic stress | Week 0, 6 and 12
  Chronic stress measured using the Wheaton Chronic Stress Questionnaire. Individual scores range from 0 to 102, with higher scores indicating higher chronic stress.
Change in self-reported sleep quality | Week 0, 6 and 12
  Sleep quality assessed by self-report using the Pittsburgh Sleep Quality Index
Change in mood | Week 0, 6 and 12
  Mood assessed using the Profile of Mood States (POMS) Standard Score. Total Mood Disturbance (TMD) score is found from the difference between "negative" subscales - "positive" subscales. Individual scores on the POMS range from -32 to 200 with higher scores indicating higher mood disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No